CLINICAL TRIAL: NCT00415896
Title: Impact of Respiratory Muscle Unloading on Respiratory Muscle Endurance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Krankenhaus Kloster Grafschaft (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: FKKG3
Record Dates: First submitted 2006-12-22; First posted 2006-12-25 (Estimated); Last update posted 2006-12-25 (Estimated); Status verified 2006-12

CONDITIONS: Chronic Respiratory Failure
Keywords: weaning; work of breathing; spontaneous breathing trial; rapid shallow breathing
MeSH Terms: interventions — Positive-Pressure Respiration

INTERVENTIONS:
Device: positive pressure ventilation

SUMMARY:
This study investigates how different degrees of muscular unloading during mechanical ventilation impact endurance of succeeding spontaneous breathing trials

DETAILED DESCRIPTION:
Liberation from mechanical ventilation in difficult to wean patients is best accomplished by intermittent spontaneous breathing trials (1). Optimal respiratory muscle rest in-between breathing trials however has never been investigated.

Using a crossover design, patients are to be ventilated with complete and partial respiratory muscle unloading for a period of ten hours respectively. Respiratory muscle activity is being monitored by oesophageal balloon technique using a commercially available System (Avea, Viasys, Conshohocken, PA, USA). Time of spontaneous breathing, respiratory- and ABG parameters are being determined to characterize the course of each spontaneous breathing trial.

References

1. Esteban, A., F. Frutos, M. J. Tobin, I. Alia, J. F. Solsona, I. Valverdu, R. Fernandez, M. A. de la Cal, S. Benito, R. Tomas, and et al. 1995. A comparison of four methods of weaning patients from mechanical ventilation. Spanish Lung Failure Collaborative Group. N Engl J Med 332(6):345-50.

ELIGIBILITY:
Inclusion Criteria:

* hypercapnic respiratory failure

Exclusion Criteria:

* upper Gi pathology
* renal failure (creatinin > 2 mg/dl)
* Sepsis or infection
* age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2006-12; Study Completion 2007-06

PRIMARY OUTCOMES:
Endurance time

SECONDARY OUTCOMES:
PCO2, respiratory parameters

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Dellweg, M.D., Principal Investigator — FKKG; Dieter Koehler, M.D., Prof., Study Chair — FKKG
Locations (1):
- Kloster Grafschaft, Schmallenberg, Annostr. 1, Germany